CLINICAL TRIAL: NCT01645319
Title: A Prospective Observational Study Comparing the Effectiveness of Treatment Strategies for Open-Angle Glaucoma
Brief Title: Comparative Effectiveness of Treatment Strategies for Primary Open-Angle Glaucoma
Acronym: RiGOR
Status: Completed | Type: Observational
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: American Academy of Ophthalmology (Other); Jules Stein Eye Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HHSA29020050035I
Record Dates: First submitted 2011-10-20; First posted 2012-07-20 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2012-07

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (12):
- White, non-hispanic - Medication Treatment Pathway
- White, non-Hispanic - Laser Surgery Treatment Pathway
- White, non-Hispanic - Incisional/Other Treatment Pathway
- Hispanic - Medication Treatment Pathway
- Hispanic - Laser Surgery Treatment Pathway
- Hispanic - Incisional/Other Surgery Treatment Pathway
- Asian - Medication Treatment Pathway
- Asian - Laser Surgery Treatment Pathway
- Asian - Incisional/Other Surgery Treatment Pathway
- Black - Medication Treatment Pathway
- Black - Laser Surgery Treatment Pathway
- Black - Incisional/Other Surgery Treatment Pathway

SUMMARY:
The primary objectives of the study are:

1. To compare the proportion of patients who achieve a successful response to treatment (reduction in Intraocular Pressure (IOP) of >15%) between patients treated with laser surgery (including argon laser trabeculectomy, and selective laser trabeculoplasty) with patients receiving additional medications, at 1-year post-treatment initiation.
2. To compare the proportion of patients who achieve a successful response to treatment (reduction in IOP of >15%) between patients treated with other procedures (including incisional surgery, drainage device procedures, and other glaucoma procedures) with patients receiving additional medications, at 1-year-post-treatment initiation.

The study is a prospective, observational cohort study and will not provide or recommend any treatment. Patients who have failed initial medical therapy with two glaucoma medications will be identified and enrolled at the time of scheduling of a laser surgery procedure or other procedure such as incisional surgery or drainage device, or initiation of an additional course of therapy with medication as determined by their physician. This inception cohort of new initiators of laser surgical treatment, other procedures, or additional medical therapy will be followed for 12 months. All decisions regarding treatment are solely at the discretion of the physician in accordance with their usual practice. Enrollment is expected to begin in February 2011 and continue through 12 months of follow-up after enrollment targets have been reached.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with open-angle glaucoma who have a new or change in therapy (decision to proceed to laser or incisional surgery or initiate a new or additional course of medication).
* Includes patients with normal-tension glaucoma, pigmentary glaucoma and pseudoexfoliation.
* Patients willing to complete visual function and quality of life questionnaires

Exclusion Criteria:

* Patients currently treated with four or more glaucoma medications (at time of enrollment).
* Patients with no light perception, or otherwise not eligible for further treatment
* Patients who have neovascular glaucoma, patients with uveitis-associated glaucoma, or patients with angle recession glaucoma.
* Patients with primary angle-closure or secondary angle-closure glaucoma
* Patients who have had prior incisional surgery for glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the United States, the prevalence of open-angle glaucoma for all adults 40 years old and older is estimated to be 1.86%. Open-angle glaucoma affects an estimated 2.22 million people, and that will rise to 3.3 million in 2020 as the population ages in the United States. Worldwide, it is estimated that 66.8 million people have glaucoma. Glaucoma of all types is one of the leading causes of legal blindness in the country.
Sampling Method: Non-Probability Sample
Enrollment: 2597 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary outcomes of interest are IOP, visual function, and quality of life. | 12 Months

SECONDARY OUTCOMES:
Secondary outcomes of interest include visual field assessment, visual acuity, treatment complications and repeat surgeries. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Rich Gliklich, MD, Principal Investigator — Outcome DEcIDE Center
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States